CLINICAL TRIAL: NCT05481658
Title: A Phase I, Open Label Study Employing the Topical Immunomodulator Diphencyprone to Improve Efficacy of PD-1 or PD-L1 Immune Checkpoint Inhibition in the Treatment of Advanced Cancer With Cutaneous Metastases
Brief Title: Diphencyprone Plus Immune Checkpoint Inhibition in the Treatment of Cutaneous Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nicholas Gulati (Other)
Responsible Party: Sponsor-Investigator, Nicholas Gulati, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-01421
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cutaneous Metastases
MeSH Terms: interventions — diphenylcyclopropenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diphencyprone (DPCP) (Experimental): 0.4% and 0.04% ointment
  Interventions: Drug: Diphencyprone (DPCP)

INTERVENTIONS:
Drug: Diphencyprone (DPCP) — topical immunomodulator
  Other Names: diphencyprone

SUMMARY:
This is a phase I, open label study employing diphencyprone (DPCP) to characterize gene expression changes of various immune cell and tumor markers in cutaneous metastases treated with topical DPCP twice weekly for 12 weeks in combination with PD-1 or PD-L1 immune checkpoint inhibition (ICI), compared to pre-treatment cutaneous metastases and to describe the adverse events associated with DPCP when administered topically twice weekly for 12 weeks in combination with PD-1 or PD-L1 ICI.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed cancer with at least three cutaneous metastasis sites that are able to be biopsied.
* Subject's oncologist plans as next standard of care treatment to use an FDA- approved PD-1 or PD-L1 ICI therapy. In other words, the subject would be treated with PD-1 or PD-L1 ICI therapy even if not taking part in this study. Subjects can be either ICI-naïve (never having received ICI previously), or may have progressed/relapsed during ICI therapy, but the treating oncologist has elected to continue PD-1 or PD-L1 ICI therapy.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately:
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Subjects may not be receiving any other investigational agents.
* Subjects must not be receiving combination ICI, such as a PD-1 inhibitor with a CTLA-4 inhibitor.
* Subjects taking any of the following systemic therapies: corticosteroids, immunosuppressants, and/or any other medications (systemic or topical) that may affect the outcome of the study in the opinion of the investigator
* Subjects with any underlying diseases or dermatological conditions of the affected areas that require the use of interfering topical or systemic therapy, or that may, in the opinion of the investigator, impair immune responses such as HIV or lymphadenectomy of the axillary lymph node basin that drains the skin where DPCP is to be applied.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to DPCP, or any of the other components of the DPCP ointment formulation.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with a grade 3 adverse event | at Day 98 or 128
  Safety and tolerability of dual-therapy DPCP plus immune checkpoint inhibition will be measured as the proportion of subjects with a grade 3 on the Common Terminology Criteria for Adverse Events (CTCAE) criteria for eczema, version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Gulati, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Philip Friedlander, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  Any purpose. Specify Other Mechanism PI to be contacted